CLINICAL TRIAL: NCT02492919
Title: Impact of Medixair® System on Surgical Site Infection in Patients Admitted Into the Postoperative Cardiac Intensive Care Unit
Brief Title: Medixair® System on Surgical Site Infection in Cardiac Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valladolid (Other)
Collaborators: Hospital Clínico Universitario de Valladolid (Other)
Responsible Party: Principal Investigator, F. Javier Alvarez, Professor, University of Valladolid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PI 14-176; 17-01-2011 (Other: Comision Investigacion HCUV)
Record Dates: First submitted 2015-05-04; First posted 2015-07-09 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Surgical Site Infection
Keywords: cardiac surgery; risk factors; infection
MeSH Terms: conditions — Surgical Wound Infection; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medixair® (Experimental): Cardiac reanimation unit bed with Medixair®
  Interventions: Device: Medixair®
- NO Medixair® (No Intervention): Cardiac reanimation unit bed with NO Medixair®

INTERVENTIONS:
Device: Medixair® — Medixair system uses C-ultraviolet rays, which are the strongest ultraviolet kind of rays to kill microorganisms. The intervention consist consists of adding the Medixair® device, to be various beds of Cardiac Reanimation Units, or not.
  Arms: Medixair®

SUMMARY:
There is a growing incidence of sepsis and septic shock in people after surgery, for which there may be several reasons: more elderly people and more severe illnesses are entering operating theatres, more invasive systems are being used to take care of patients in intensive care units, etc... Sepsis and septic shock are the most prevalent illnesses which cause the highest mortality in intensive care units.

The incidence of this illness is 500,000 / year in the USA, and 240-400 / 100,000 persons in Europe. So this is a subject of great interest in hospitals and also to the National Health System (to both health workers and the health authorities) as a lot of money is spent on this illness.

Since the 19th century, ultraviolet rays have been known to be able to sterilize microorganisms (to kill them); yet no ultraviolet system machine has been on the market, until now, to control nosocomial infections.

The Medixair system, which aims to do this, has recently come on to the market. It uses C-ultraviolet rays, which are the strongest kind of ultraviolet rays to kill microorganisms.

Thus, it is of interest to know whether this system is good enough to lower infections in intensive care units. It is logical to believe that the the fewer the micro-organisms, the lower the possibilities of infection.

DETAILED DESCRIPTION:
Study design Prospective, comparative, randomized, non intervention study

Patients

Patients older than 18 years

Cardiac Surgery anesthetized using Extracorporeal Circulation

Randomization

There are 10 independent boxes at the Postoperative Cardiac Intensive Care Unit. (Each of these boxes have single beds). Every year, the Cardiac Reanimation Unit of our hospital received 500 patients, post heart surgery.

After getting the permissions needed to make the research, the Medixair® system has been placed in 5 of these units, and the comparison group will be the other 5 beds without Medixair®. Patients have been assigned randomly to either (Medixair® and NO Medixair®).

The endpoint is:

-To compare the infection rates after a cardiac surgery, on patients located in boxes with and without a Medixair® system.

The aim is to see if there are fewer catheter infections, less bacteraemia, fewer urinary infections, less site of surgery infections, and fewer pneumonias in patients who have spent their first days after a heart surgery in a box with Medixair® system than without it. The infection rates in the intensive care unit will be followed, as well as the whole stay at hospital, as there might be fewer infections if there were fewer microorganisms around.

Other objectives are:

* Identifying preoperative, intraoperative and postoperative risk factors to develop an infection illness after cardiac surgery, as well as which increase the length of stay at hospital and the mortality rate.
* Making an economic study of using this system against not using it.

A further aim is to measure the following variables:

* Dependent variables (Outcome variables): infection
* 2º Outcome variables: colonization
* Independent variables will be a risk factor for infection:
* Preoperative: age, sex, any preoperative illness, immunosuppressor treatment, including corticosteroids.
* Intraoperative: antibiotic prophylaxis, surgical technique, length of cardiopulmonary bypass, length of aorta clamped, temperature during cardiopulmonary bypass, hematocrit at the end of cardiopulmonary bypass.
* Postoperative: length with mechanical ventilation, time spent in hospital, time spent in an intensive care unit, any organ complication (pulmonary insufficiency, renal failure, low cardiac index), septicemia, invasive techniques used, positive microorganism cultures.

All of the patients will be treated in the same way

Estimated number of patients

Nowadays, the infection rate after cardiac surgery is around 5%, so following the current hypothesis that the Medixair® system, because of its ultraviolet emissions, is going to lower the infection rate after cardiac surgery, 419 patients are needed in each group to be able to demonstrate a significative 5% reduction in infection rates, with an alpha error of 0.05 and a beta error of 0.2 to have a power of 80%.

As this is a preliminary study, in order to demonstrate a 5% reduction in the infection rate, half the number of patients (half of 419) will be used. As the patient volume is 500 a year, the number will be rounded up to 500, in order to be able to consider a complete year.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to Postoperative Cardiac Intensive Care Unit after Cardiac Surgery with Extracorporeal Circulation

Exclusion Criteria:

* Not signing informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2011-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Infection rates after cardiac surgery | 3 weeks
  To assess if there are fewer catheter infections, less bacteraemia, fewer urinary infections, fewer surgery site infections, fewer pneumonias in patients who have spent their first days after a heart surgery in a box with the Medixair system than without it.

SECONDARY OUTCOMES:
Number of infected patients | 3 weeks
  Number of infected patients
mortality rate | 3 weeks and for the whole stay at hospital
  mortality rate
number of patients with pneumonia | 3 weeks
  number of patients with pneumonia

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Tamayo, PhD, MD, Study Director — Hospital Clínico Universitario de Valladolid